CLINICAL TRIAL: NCT04712656
Title: Effects of CPAP Therapy on Blood Pressure and Heart Rate Variability in Obstructive Sleep Apnea: Role of Symptom Subtypes
Brief Title: Effects of CPAP Therapy on Blood Pressure and Heart Rate Variability in Obstructive Sleep Apnea
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: University of Pennsylvania (Other); Chang Gung Memorial Hospital (Other); University of Sydney (Other); The University of Western Australia (Other); Peking University (Other); Ruijin Hospital (Other); National University of Singapore (Other); University of Iceland (Other); Geisinger Health (Unknown); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Ulysses Magalang MD, Professor of Internal Medicine, Ohio State University
Other Study IDs: 2020H0524
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Cardiovascular
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- OSA Subjects Treated with CPAP: Patients with moderate to severe OSA (ODI4>15/h) who accept CPAP therapy.
  Interventions: Device: CPAP therapy

INTERVENTIONS:
Device: CPAP therapy — CPAP treatment of obstructive sleep apnea.

SUMMARY:
The primary objective of this study is to determine whether the effect of continuous positive airway pressure (CPAP) therapy on 24-hour mean blood pressure (BP) in patients with obstructive sleep apnea (OSA) varies between symptom phenotypes.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, multi-center, cohort study involving patients with moderate to severe OSA. This study will compare OSA patients who accept and comply with CPAP therapy versus those who do not.

Variables of Interest: 24-hour ambulatory BP, sitting BP, electrocardiogram (ECG), facial photographs, psychomotor vigilance test (PVT), questionnaires, and blood samples.

Patients will complete questionnaires that pertain to demographics, lifestyle factors, and co-morbidities associated with CVD. The blood samples will be used to look for evidence of diabetes; elevated lipids; markers of heart injury, inflammation, and coagulation; and genetic information. Measurements will be collected at baseline and at 6-month follow-up.

In addition, patients enrolled in this study will be contacted by telephone once a year over a ten year period. The purpose of the telephone interview is to determine if they are using any treatment for OSA, if they have developed any new health problems such as a heart attack or stroke, and if they have changed any of their usual medications.

Data Analysis Approach: To correct for potential bias in the non-randomized comparison, we will apply a Propensity Score (PS) Design via subclassification. Models to derive the PS values used in this design will include a number of covariates relevant to CPAP adherence and cardiovascular outcomes, including age, sex, obesity (BMI, neck circumference, waist-to-hip ratio), current smoking, prevalent CVD at baseline, history of hypertension, HbA1c, diabetes mellitus (history, medications), lipid profile, hyperlipidemia (history, medications), family history of premature coronary disease, Charlson comorbidity index, physical activity (IPAQ), diet, OSA severity (AHI, ODI4, T90), sleepiness (Epworth Sleepiness Scale), educational attainment, socioeconomic status (postcode), insomnia symptoms (Insomnia Symptom Questionnaire), anxiety and depression-related symptoms (Patient Health Questionnaire-2), self-efficacy (General self-efficacy scale), and medication adherence (Medication Adherence Report Scale [MARS-5]). Baseline values of outcome measures will also be included in the PS model. After creating the PS design, all analyses are performed accounting for PS subclass as a categorical stratification factor. Evaluations of the CPAP effect on binary outcomes are performed utilizing conditional logistic regression. Similarly, CPAP effects in the context of survival analyses (e.g., Cox Proportional Hazards models) or on continuous outcomes (e.g., linear regression) are assessed by including PS subclass as a categorical covariate in all models.

ELIGIBILITY:
Inclusion Criteria:

* 30 to 75 years of age
* Among patients with hypertension, no change in BP medication for at least 3 months.
* Willing and able to give informed consent
* Willing and able to complete ambulatory blood pressure monitoring at baseline and after 6-months.
* Sleep study [Polysomnography (PSG) or Home Sleep Apnea Study (HSAT) performed based on clinical grounds
* 4% oxygen desaturation index (ODI4) ≥15 events/hour on clinical sleep study
* Planned CPAP treatment by treating provider

Exclusion Criteria:

* Unable to apply BP cuff (e.g. arm circumference >55 cm, prior breast cancer, structural abnormalities of the arm)
* Current use of CPAP or Dental Device for OSA
* Category III-IV of heart failure
* Presence of Cheyne-Stokes Respiration (CSR) in PSG
* Predominantly central sleep apnea (AHI≥15 events/hour)
* Pregnancy
* History of renal failure, or renal transplant
* Self-reported sleep duration less than 5 hours per night on weeknights (work nights)
* Other sleep disorders
* Use of supplemental oxygen during wakefulness or sleep
* Self-reported illicit drug use or marijuana use more than once per week
* Unstable medical conditions: uncontrolled angina, uncontrolled hypertension, severe chronic obstructive pulmonary disease, active cancer, or unstable psychiatric disease
* Any underlying condition that, in the opinion of the lead investigator, prohibits participation in the study
* Development or adoption of any of the above exclusion criteria during the study period

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults between the ages of 30 to 75 years old with moderate to severe obstructive sleep apnea (OSA). OSA diagnosis will be defined as an apnea/hypopnea index (AHI) >or =5 episodes per hour.
Sampling Method: Probability Sample
Enrollment: 1739 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2031-03-01 (Estimated); Study Completion 2032-03-01 (Estimated)

PRIMARY OUTCOMES:
24-hour Mean Blood Pressure | Measurements will be conducted at baseline (prior to CPAP therapy) and 6-months after initiation of CPAP therapy.
  24-hour Mean Blood Pressure obtained from ambulatory blood pressure monitoring (ABPM)

SECONDARY OUTCOMES:
Heart Rate Variability | Measurements will be conducted at baseline (prior to CPAP therapy) and 6-months after initiation of CPAP therapy.
  Heart Rate Variability obtained from 5-minute ECG

CONTACTS AND LOCATIONS:
Overall Officials: Ulysses Magalang, MD, Principal Investigator — Ohio State University
Locations (1):
- Martha Morehouse Medical Pavilion, Suite 2600, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No